CLINICAL TRIAL: NCT01274858
Title: Sensory Mapping and Thermal Thresholds After Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H-B-2008-059/6
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-02

CONDITIONS: Lung Cancer
Keywords: persistent pain; neuropathic pain; Thoracotomy; Chronic Pain
MeSH Terms: conditions — Lung Neoplasms; Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung cancer surgery

SUMMARY:
The study will investigate topography of sensory changes late after lung cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* Understand Danish
* Age > 18 years old
* PTPS

Exclusion Criteria:

* Cognitive dysfunction
* Repeated thoracic surgery
* Nerve injury from other causes
* Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Thermal thresholds (Quantitative Sensory Testing [QST]) | average 18 months after surgery
  Two QST with 10 days interval
Sensory mapping | average 18 months after surgery
  Two QST with 10 days interval

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Section for Surgical Pathophysiology 4074, Copenhagen

REFERENCES:
- [Derived] Werner MU, Ringsted TK, Kehlet H, Wildgaard K. Sensory testing in patients with postthoracotomy pain syndrome: Part 1: mirror-image sensory dysfunction. Clin J Pain. 2013 Sep;29(9):775-83. doi: 10.1097/AJP.0b013e318277b646. PMID 23328340